CLINICAL TRIAL: NCT07132346
Title: "Are Women Hesitant to Become Mothers in the New World?"
Brief Title: Are Women Hesitant to Become Mothers in the New World?
Acronym: aging
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Ece Kaplan, Asst. Prof., University of Gaziantep
Other Study IDs: GAUN-EBE-EKD-02; UGaziantep (Registry Identifier: ECE KAPLAN)
Record Dates: First submitted 2025-07-23; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Women (Between 18 to 50 Years Old)
Keywords: maternal ambivalence; avoiding pregnancy; women; aging anxiety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AGING ANXIETY SCALE — This study was conducted as descriptive research to determine the mediating role of aging anxiety in the relationship between maternal ambivalence and pregnancy avoidance in women.

SUMMARY:
The decision to have a child can be perceived as indecisive, and women who experience maternal indecisiveness avoid pregnancy. However, as women age, fertility anxiety also increases. The investigators aimed to investigate the mediating role of aging anxiety in the relationship between maternal ambivalence and avoidance of pregnancy in women.

DETAILED DESCRIPTION:
The decision to have a child can be perceived as indecisive, and women who experience maternal indecisiveness avoid pregnancy. However, as women age, fertility anxiety also increases. We aimed to investigate the mediating role of aging anxiety in the relationship between maternal ambivalence and avoidance of pregnancy in women. Data collection tools included a "Personal Information Form," "the Maternal Ambivalence Scale," "the Desire to Avoid Pregnancy Scale," and "The Relational Aging Anxiety Scale." Regression models assessed the association between Maternal Ambivalence Scale, Desire to Avoid Pregnancy Scale and Relational Aging Anxiety Scale. SPSS Process v.3.4 analysis was performed to make a mediator effect assessment. It was found that the model was significant and 3% of the desire to avoid pregnancy was explained by maternal ambivalence (F=9.088; p=0.003) (n=300). Since the confidence interval (95% CI [0.019; 0.096]) of the indirect effect did not include "0", a mediating effect was detected. It was found that the model was significant and 17.6% of the desire to avoid pregnancy was explained by the doubts sub-dimension (F=9.477; p=0.002). Since the confidence interval (95% CI [0.024; 0.200]) of the indirect effect did not include "0", a mediating effect was identified. The collective affinity for older people sub-dimension had a partial mediating effect between rejection and the desire to avoid pregnancy. Results indicated that 20.5% of the total effect on the desire to avoid pregnancy was provided by the mediating effect. It was found that women's perceptions of aging caused maternal ambivalence and that this situation was effective in avoiding pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Having no communication barriers,
* Age ≥20 years, and
* Being married.

Exclusion Criteria:

* Unwilling to participate in the study,
* Having a psychiatric health problem according to medical records,
* Being single, and
* Being pregnant.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study consisted of women aged ≥20 years who applied to the obstetrics and gynecology clinic of XXX hospital for any reason. A literature review was conducted and a power analysis was performed on the G-power 3.9.1 software to calculate the sample size following a literature review (Guney et al., 2022; Gipson et al., 2021). The minimum sample size required to expect a significant relationship with a large effect size (Cohen's d=0.0784314) in terms of women's tendency to avoid pregnancy was found to be 300 individuals (α=0.05, 1-β=0.95). Totally, 312 women were reached, but 12 were not included in the study as they dropped out. Eventually, the study sample consisted of 300 women.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
"the Maternal Ambivalence Scale" | 3 MONTHS
  The study sample consisted of 300 women. Their written and verbal consent was obtained.
  The Maternal Ambivalence Scale: The scale has 14 four-point Likert-type items, each of which is scored between 1 and 4. The minimum total score that can be obtained from the scale is 14, and the maximum is 56. An increase in the total score indicates a high level of maternal ambivalence. The scale has three sub-dimensions.
The Desire to Avoid Pregnancy Scale | 3 months
  The Desire to Avoid Pregnancy Scale: The five-point Likert-type items on the scale are scored using the following options: "0= strongly agree" and "4= strongly disagree. Scores on the scale range from 0/14=0 to 56/14=4. A high score obtained from the scale indicates an increase in the desire to avoid pregnancy, while a low score shows a decrease in this respect.
The Relational Aging Anxiety Scale | 3 months
  The Relational Aging Anxiety Scale: Items are scored on a five-point Likert-type scale from (1) strongly agree to (5) strongly disagree. The scale consists of three sub-dimensions. The scale does not have a total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Development and psychometric properties of the maternal ambivalence scale in spanish women — https://bmcpregnancychildbirth.biomedcentral.com/articles/10.1186/s12884-022-04956-w